CLINICAL TRIAL: NCT03643341
Title: Family-based, Healthy Living Intervention for Children With Overweight and Obesity and Their Families
Brief Title: Family Healthy Living Early Intervention Program
Acronym: EIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Victoria (Other)
Collaborators: Childhood Obesity Foundation (Other)
Responsible Party: Principal Investigator, Patti-Jean Naylor, Professor, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BC18-024
Record Dates: First submitted 2018-07-06; First posted 2018-08-22 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Health Behavior; Child Behavior; Child Obesity; Nutrition Disorders; Body Weight
Keywords: Family-based; Community-based; Healthy Weights
MeSH Terms: conditions — Obesity; Health Behavior; Child Behavior; Pediatric Obesity; Nutrition Disorders; Body Weight

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Healthy Living Intervention (Experimental): Children aged 8-12 and at least one caregiver will meet for 10 weekly face-to-face and online intervention sessions (1.5 hours per session). Four biweekly maintenance sessions will follow the main program.
  Interventions: Behavioral: Family Healthy Living
- Wait-list control group (No Intervention): Children aged 8-12 will be randomly assigned to the wait-list control group until after the study.

INTERVENTIONS:
Behavioral: Family Healthy Living — Children aged 8-12 and at least one caregiver will meet for 10 weekly intervention sessions (1.5 hours per session), and 4 extra sessions to be chosen by families and intervention Leaders. During the intervention, participants will also have access to digital educational content that is supplementary to what is provided during the individual sessions. Four biweekly maintenance sessions will follow the main program.
  Arms: Family Healthy Living Intervention

SUMMARY:
The Childhood Healthy Weights Early Intervention Program (EIP) is a family-based pilot program that will promote healthy lifestyle practices for families whose children are off the healthy weight trajectory (e.g., BMI ≥ 85th percentile for age and sex) that do not need the intensive services of medically supervised programs. It is a lifestyle behaviour approach for promoting healthy weights in children. The EIP program consists of 10 weekly intervention sessions (1.5 hours per session) followed by 4 maintenance sessions and is age specific (age 8-12). During the intervention, participants will also have access to digital educational content that is supplementary to what is provided during the individual sessions. The program will be integrated and aligned with existing BC-specific childhood healthy weights programs (e.g. the HealthLinkBC Eating and Activity Program for Kids). The EIP pilot will run from October-December 2018 with 8 child programs (age 8-12). Participants who do not qualify for this program (e.g., BMI ≤ 85th percentile for age and sex) will be offered a 10 week online program which is similar in educational content as the EIP program.

ELIGIBILITY:
Inclusion Criteria:

* Child with BMI ≥ 85th percentile for age and sex
* Child is accompanied by a parent or legal guardian
* At least one member of the family have to be able to speak and read English
* Family agrees to attend group meetings over 10 weeks

Exclusion Criteria:

* Child unavailable to attend group weekly sessions
* Parent or guardian unavailable to attend group weekly sessions
* Participating child or parent, according to parent report, has medical condition contraindicating mild energy restriction or moderate physical activity, and medical clearance was not obtained

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2018-10-10 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in BMI calculated from measures of height and weight | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Measures of height and weight will be obtained from all children. BMI will be calculated as weight (kilograms) divided by height (meters) squared, adjusted for child age and sex.

SECONDARY OUTCOMES:
Changes in BMI z-score calculated from measures of height and weight | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Measures of height and weight will be obtained from all children, BMI z-scores (standard deviation) will be calculated.
Changes in Physical Activity Engagement assessed by the Physical Activity Questionnaire for Children (PAQ-C) | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Self-reported child usual physical activity engagement will be assessed by PAQ-C 7-day physical activity recall
Changes in Physical Activity Motivation and Confidence assessed by the Canadian Assessment of Physical Literacy (CAPL-2) Physical Activity Motivation and Confidence subscale | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. The Motivation and Confidence sub-scale of CAPL-2 assesses physical activity predilection and adequacy, perceived physical activity intrinsic motivation and competence
Changes in Physical Activity assessed by the PACE Adolescent Psychosocial Measures | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. The PACE Adolescent Psychosocial Measures assesses physical activity, confidence, and family support
Changes in Sedentary Habits assessed by the PACE Adolescent Psychosocial Measures | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. The PACE Adolescent Psychosocial Measures assesses sedentary habits, confidence, and family support
Changes in Fundamental Movement Skills (FMS) assessed by the Canadian Agility and Movement Skill Assessment (CAMSA) | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  CAMSA is the FMS course from the Canadian Assessment of Physical Literacy (CAPL-2) that assesses two-foot jumping, sliding, catch, throw, skip, one-foot hop, and kick. Children will observe two demonstrations, will complete two trials, and two timed and scored trials.
Changes in Dietary Behaviours assessed by the LiGHT questionnaire (7-day recall questions retrieved from CDC BRFSS surveys) | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. Dietary behaviours such as fruits, vegetables, fruit juice, soda, fruit-flavored beverages, and pastries intake will be assessed by the 7-day dietary recall
Healthy Eating Outcome Expectations assessed by the Power Play! Survey. | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. Knowledge or ideas about what will happen when regularly consuming fruits and vegetables.
Changes in Dietary Behaviors Self-efficacy assessed by the PACE Adolescent Psychosocial Measures | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. Self-efficacy to increase fruit and vegetable intake, and to reduce the intake of sugary beverages and sweet/salty snack foods will be assessed.
Changes in Healthy Eating Motivation assessed by the FLASHE questionnaire | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. Motivation for eating fruits and vegetables will be assessed. Motivation for limiting sweet/salty snack foods and sugary drinks will also be assessed.
Changes in Perceived Cooking Skill assessed by the Cooking with Kids questionnaire | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. Assesses child's ability to prepare and cook food
Changes in Self-esteem assessed by the Project EAT survey | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. Self-esteem will be assessed by the Project EAT survey
Changes in Gratitude assessed by the Gratitude Adjective Checklist | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. Changes in Gratitude assessed using the Gratitude Adjective Checklist
Changes in Self-compassion by the Self-compassion Scale Short Form | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. Changes in Gratitude assessed using the Self-compassion Scale Short Form
Changes in Sleep Habits assessed by the FLASHE questionnaire | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Child questionnaire. Usual hours of sleep will be self-reported by the child
Changes in Parent Feeding Practices assessed by questions drawn from the FLASHES-EAT surveys. | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. The FLASHES-EAT survey assess how parents communicate with their children regarding food and dietary habits and how they organize and monitor the home food environment.
Changes in Parent Feeding Practices assessed by a question drawn from the CANPOWER questionnaire | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. The CANPOWER questionnaire assesses whether or not parents encourage their child to participate in healthy lifestyle behaviors (eating fruits and vegetables)
Changes in Parent Feeding Practices assessed by the Parent Support of Healthy Eating questionnaire | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. This questionnaire assess each parent's specific behavioral constructs (affective attitude, instrumental attitude) in regards to supporting their child's healthy eating behaviors.
Changes in Structure of the Home Food Environment assessed by the Fruit and Vegetable At Home Survey For Parents. | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. The Fruit and Vegetable At Home Survey For Parents assess the availability and accessibility of fruits and vegetables within the home.
Changes in Parent's Personal Dietary Behaviours are assessed by the FLASHE questionnaire. | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. The FLASHE questionnaire assess parents' fruit and vegetable intake in addition to their consumption of food away from the home (e.g. fast-food restaurants, work cafeteria).
Changes in Parent Food Preparation Self-efficacy assessed with two questions drawn from the FLASHES-EAT survey. | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. The questions drawn from the FLASHES-EAT survey assess parents' confidence level with preparing a variety of fruits and vegetables as well as their level of confidence preparing family meals with their children.
Changes in Behavioral Regulation of Supporting Child's Healthy Eating assessed by the Action Control of Parent Support Behaviour | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. This questionnaire assess whether or not parents set goals and make regular plans to support their child's healthy eating behaviors.
Changes in Healthy Eating Habits assessed by the automaticity subscale of Self-Report Index of Habit. | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. The Self-Report Index of Habit assess whether or not parents believe that preparing and eating healthy meals is something their family does habitually.
Changes in Healthy Eating Identity assessed by the Role-Identity subscale from the Exercise Identity Scale. | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. These questions assess how parents view their own and their family's dietary behaviors and food choices.
Changes in Parent Physical Activity Support assessed by the ParticipACTION 24hr Guidelines Survey | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. Changes in Parent Physical Activity Support will be assessed by the ParticipACTION 24hr Guidelines Survey
Changes in Parent Physical Activity Self-efficacy assessed by the LiGHT study questionnaire | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. Changes in Parent Physical Activity Self-efficacy assessed by the LiGHT study questionnaire
Changes in Behavioral Regulation of Supporting Child's Physical Activity assessed by the Action Control of Parent Support Behaviour | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. This questionnaire assess whether or not parents set goals and make regular plans to support their child's physical activity participation.
Changes in Physical Activity Habit assessed by the automaticity subscale of the Self-Report Index of Habit | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. The Self-Report Index of Habit assess whether or not parents believe that participating in physical activity is something their family does habitually.
Changes in Physical Activity Identity assessed by the Role-Identity subscale from the Exercise Identity Scale. | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. These questions assess how parents view their own and their family's physical activity participation.
Changes in Parent Support for Child Sleep Habits assessed by the ParticipACTION 24hr Guidelines Survey | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. Changes in Parent Support for Child Sleep Habits will be assessed by the ParticipACTION 24hr Guidelines Survey
Changes in Child Quality of Life assessed by the Pediatric Quality of Life Inventory | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Parent questionnaire. Changes in Child Quality of Life will be assessed by the Pediatric Quality of Life Inventory

OTHER OUTCOMES:
Process Evaluation of the EIP | Baseline, post-intervention (10 weeks), and post-maintenance (18 weeks)
  Evaluate the reach, implementation, and sustainability of the EIP. Examine if the EIP is reaching a broad demographic, if families and staff are satisfied with the EIP, if the EIP is being implemented as intended across the pilot sites and to explore the facilitators and barriers to implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Strange, PhD, Study Director — Childhood Obesity Foundation
Locations (10):
- Canada (10):
  - Cameron Recreation Centre, Burnaby, British Columbia
  - Strathcona Gardens Recreation Complex, Campbell River, British Columbia
  - Neighbourhood Learning Centre, Chilliwack, British Columbia
  - Kelowna Family YMCA, Kelowna, British Columbia
  - Cowichan Open Learning/Duncan Elementary School, North Cowichan, British Columbia
  - YMCA Northern BC, Prince George, British Columbia
  - Tong Louie YMCA, Surrey, British Columbia
  - Surrey Sport & Leisure Complex, Surrey, British Columbia
  - Langara Family YMCA, Vancouver, British Columbia
  - Juan de Fuca Recreation Centre, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be share with co-investigators

REFERENCES:
- [Derived] Perdew M, Liu S, Rhodes R, Ball GDC, Masse LC, Hartrick T, Strange K, Naylor PJ. The Effectiveness of a Blended In-Person and Online Family-Based Childhood Obesity Management Program. Child Obes. 2021 Jan;17(1):58-67. doi: 10.1089/chi.2020.0236. Epub 2020 Dec 23. PMID 33370164
- [Derived] Liu S, Marques IG, Perdew MA, Strange K, Hartrick T, Weismiller J, Ball GDC, Masse LC, Rhodes R, Naylor PJ. Family-based, healthy living intervention for children with overweight and obesity and their families: a 'real world' trial protocol using a randomised wait list control design. BMJ Open. 2019 Oct 31;9(10):e027183. doi: 10.1136/bmjopen-2018-027183. PMID 31676642